CLINICAL TRIAL: NCT07029009
Title: Investigating Enteroendocrine Dysfunction, Metabolism, and Response to Liraglutide in Patients With Maturity-onset Diabetes of the Young (MODY)
Brief Title: Liraglutide Treatment in Patients With Maturity-onset Diabetes of the Young (MODY)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mansa (Other)
Responsible Party: Sponsor-Investigator, Mansa, ASSISTANT PROFESSOR, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0426
Record Dates: First submitted 2024-08-19; First posted 2025-06-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2024-12

CONDITIONS: Maturity Onset Diabetes of the Young
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- liraglutide treatment (Experimental): After baseline evaluation of enteroendocrine levels and metabolism, study participants will be prescribed liraglutide. Titration of liraglutide will be as follows: 1) Starting dose of liraglutide 0.6 mg daily for 1 week, 2) Increase to liraglutide 1.2 mg daily for 1 week, and 3) Maintain at final dose of liraglutide 1.8 mg daily. If study participants are unable to tolerate liragultide 1.8 mg daily due to side effects for 1 week, then will decrease back to liraglutide 1.2 mg daily.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Liraglutide will be prescribed following FDA approved packet insert for type 2 diabetes in our test population.
  Other Names: Victoza; Saxenda

SUMMARY:
The reason for this research study is to better understand the use of liraglutide, a commonly prescribed Type 2 diabetes medication, in patients with a diagnosis of maturity-onset diabetes of the young (MODY).

The investigators are interested in better understanding the way that this drug affects the metabolism and hormone levels of a person with MODY. Many people with MODY report having gastrointestinal (GI) issues such as an upset stomach. Investigators also are interested in finding out if this drug will help with GI issues.

If liraglutide does help with this symptom of MODY, the investigators want to know why this happens. If this drug is effective for participants, the investigators will use participants cells to make human induced pluripotent stem cell (iPSC). This means that the investigators will use participant cells to create what are called stem cells, which are cells in the body that are able to be told what their job is. Investigators will use these cells to see what happens in gastrointestinal (GI) tract.

DETAILED DESCRIPTION:
The objective of this study is to perform a comprehensive metabolic and hormonal evaluation of individuals with Maturity-onset diabetes of the young (MODY) at baseline and then assess response to initiation of liraglutide. Select individuals will be consented for human induced pluripotent stem cell (iPSC) generation to identify the cellular basis of enteroendocrine cell (EEC) dysfunction.

The hypothesis is that heterozygous mutations in MODY-related genes contribute to a range of GI pathologies, including regional disruptions in epithelial identity and disturbances in the function of EECs. Thus, patients with MODY may experience improvement not only in HbA1c and BMI but also in GI symptoms with initiation of GLP-1 receptor agonists. Investigators plan to enroll approximately 50 patients with MODY and obtain baseline metabolic labs and imaging along with enteroendocrine labs before initiating liraglutide and assessing response with repeat labs and imaging. This project will provide further guidance for clinical care and treatment of patients with MODY.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MODY via genetic testing
* HgbA1c >6.5%

Exclusion Criteria:

* History of anaphylaxis to GLP-1 receptor agonists
* Already taking GLP-1 receptor agonists
* on medications within the stimulant class
* have had bariatric surgery
* personal or family history of cancer, especially medullary thyroid cancer
* personal history of pancreatitis or pathogenic variants associated with increased risk of pancreatitis
* known active kidney disease
* severe hypoglycemia (glucose < 50 mg/dL) within 3 months of study enrollment
* HbA1c > 10.0%
* episode of diabetic ketoacidosis (DKA) in the past 3 months
* are currently pregnant
* BMI < 18.5 kg/m2 and pediatric patients with BMI < 5th percentile

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Blood sugar control - HbA1C | Baseline and 3 months after study treatment initiation
  Hemoglobin A1c
BMI | baseline, 1 month, 2 months, and final study visit 3 months after study treatment initiation
  Body mass index; weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Metabolic - Blood Sugar | Baseline through three months of study treatment
  Glycemic patterns observed utilizing a continuous glucose monitor
Enteroendocrine function - GI symptoms | baseline, 1 month, 2 months, and final study visit 3 months after study treatment initiation
  ANMS Gastroparesis Cardinal Symptom Index Daily Diary (ANMS GCSI-DD)
Enteroendocrine function - insulin | baseline and 3 months after study treatment initiation
  Fasting and post meal blood serum insulin levels will be assessed
Enteroendocrine function - c-peptide | baseline and 3 months after study treatment initiation
  Fasting and post meal blood serum c-peptide levels will be assessed
Body fat percentage | baseline, 1 month, 2 months, and final study visit 3 months after study treatment initiation
  % body fat as identified by DXA
Liver steatosis | baseline and 3 months after treatment initiation
  MRI to determine liver health

CONTACTS AND LOCATIONS:
Overall Officials: Mansa Krishnamurthy, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be made available to other researchers.